CLINICAL TRIAL: NCT00077896
Title: Direct Current Brain Polarization in Frontotemporal Dementia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040122; 04-N-0122
Record Dates: First submitted 2004-02-12; First posted 2004-02-13 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-08

CONDITIONS: Pick Disease of the Brain
Keywords: Treatment; Transcranial Stimulation; Frontal Lobe; Pick's Disease; Cognitive Impairment; Dementia; Frontotemporal Dementia; FTD
MeSH Terms: conditions — Pick Disease of the Brain; Cognitive Dysfunction; Dementia; Frontotemporal Dementia

INTERVENTIONS:
Procedure: Direct Current Polarization

SUMMARY:
This pilot study will evaluate the effect of direct current (DC) electrical polarization of the brain on language, memory, reaction time, and mood in six patients with frontotemporal dementia (Pick's disease). There is no effective treatment available for cognitive impairment in patients with this condition. DC polarization sends a very weak current between two sponge pads placed on the head. In a previous study in healthy volunteers, DC polarization of the left prefrontal area of the brain increased verbal fluency, memory and attention, and motor reaction time in the study subjects.

Patients between 35 and 75 years of age with frontotemporal dementia who have been referred to NINDS's Cognitive Neuroscience Section for an existing protocol will be offered participation in this study. Candidates will be screened with a neurological examination to confirm the diagnosis of frontotemporal dementia.

Participants receive 40 minutes of DC polarization or sham polarization in each of two separate sessions. (No current is applied in the sham treatment). During the polarization, the patient rests quietly. Sponge pads that have been soaked in water are put on the left side of the head and above the right eye, and are held in place with elastic netting. Before the polarization and after about 20 minutes of polarization, patients undergo the following tests:

* Language: Patients must say as many words beginning with certain letters as they can in 90 seconds.
* Memory: Patients must remember a letter on a computer screen, and when the letter appears again, press the same letter on the keyboard.
* Reaction time: Patients place pegs on a pegboard.
* Mood: Patients place a mark on a line ranking how they feel.

DETAILED DESCRIPTION:
Introduction: In this study, we will use anodal direct current (DC) polarization at 2 mA to treat patients with frontotemporal dementia (FTD). Currently, there is no effective treatment for these patients. Previously, in healthy volunteers, we observed that DC polarization of the left prefrontal area for 20 min safely increases verbal fluency, cognitive processing speed (working memory and attention) and motor reaction speed. Both of these functions are severely impaired in FTD. Objective: We wish to see whether anodal DC polarization of the left prefrontal cortex in FTD patients leads to improvement in verbal fluency and working memory. Design: In this pilot study, we propose to treat six FTD patients for 40 min with anodal and sham DC polarization in a single-blind, crossover design. Outcome Measures: The main outcome measures will be verbal fluency and working memory. If anodal DC polarization produces clinically relevant improvements in these patients this will provide the impetus for a larger trial.

ELIGIBILITY:
INCLUSION CRITERIA:

-Six patients referred to the Cognitive Neuroscience Section, NINDS, with a clinical diagnosis of FTD confirmed here, will be selected to participate in the study.

EXCLUSION CRITERIA:

* Greater than 75 years of age.
* Presence of metal in the head other than dental hardware.
* Broken skin in the area of the stimulating electrodes.
* Any behavioral disorder that makes testing impossible.
* Children are excluded, as FTD is not a childhood illness.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6
Dates: Start 2004-02; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Agnew WF, McCreery DB. Considerations for safety in the use of extracranial stimulation for motor evoked potentials. Neurosurgery. 1987 Jan;20(1):143-7. doi: 10.1097/00006123-198701000-00030. PMID 3808255
- [Background] Antal A, Kincses TZ, Nitsche MA, Paulus W. Manipulation of phosphene thresholds by transcranial direct current stimulation in man. Exp Brain Res. 2003 Jun;150(3):375-8. doi: 10.1007/s00221-003-1459-8. Epub 2003 Apr 16. PMID 12698316
- [Background] Baudewig J, Nitsche MA, Paulus W, Frahm J. Regional modulation of BOLD MRI responses to human sensorimotor activation by transcranial direct current stimulation. Magn Reson Med. 2001 Feb;45(2):196-201. doi: 10.1002/1522-2594(200102)45:23.0.co;2-1. PMID 11180425